CLINICAL TRIAL: NCT00420459
Title: Aripiprazole in Fragile X Syndrome
Brief Title: A Prospective Open-label Study of Aripiprazole in Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0609-22
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aripiprazole (Experimental)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — All subjects will initially receive 2.5 mg/day of aripiprazole during the first week. The dosage may be increased to a maximum of 20 mg/day over 8 weeks.
  Other Names: Abilify

SUMMARY:
The purpose of this study is to determine the effectiveness and tolerability of aripiprazole in the treatment of children and adolescents with Fragile X Syndrome.

DETAILED DESCRIPTION:
This 12-week prospective, open-label study design was chosen to gather pilot data for potential future lager scale, double-blind, placebo-controlled studies in Fragile X Syndrome.

We hypothesize that aripiprazole will be effective in decreasing aggression, SIB, agitation, and interfering repetitive behavior commonly observed in individuals with Fragile X Syndrome. We also hypothesize that aripiprazole will be well tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 5 and 35 years and
2. Body weight greater than or equal to 15 kg
3. Confirmed diagnosis of Fragile X Syndrome based upon genetic testing results.
4. Outpatients.
5. Psychotropic medication-free for at least 2 weeks prior to screening laboratory tests and electrocardiogram. (Except 5 weeks for fluoxetine and 4 weeks for all typical and atypical antipsychotics that have been administered for at least a 4 week period.) Exceptions to medication-free status will include drugs given at bedtime targeting insomnia. Such drugs may include melatonin, clonidine, chloral hydrate, diphenhydramine, ramelteon, benzodiazepines, or other sedative-hypnotics.
6. Clinical Global Impression Scale Severity score (CGI-S) of at greater than or equal to 4 (Moderately Ill)
7. A score of at greater than or equal to 18 on the Irritability subscale of the Aberrant Behavior Checklist (ABC) at screen and baseline.
8. Mental age of greater than or equal to 18 months as measured by the Wechsler, revised Leiter, or Mullen tests
9. Each subject must be in good physical health as determined by screening procedures which will include a detailed medical history, complete physical and neurological examination.

Exclusion Criteria:

1. DSM-IV diagnosis of schizophrenia, another psychotic disorder, bipolar disorder or alcohol or other substance abuse within the last 6 months.
2. A significant medical condition such as heart, liver, renal or pulmonary disease, or an actively treated seizure disorder, as determined by history, physical examination or laboratory testing.
3. Subjects with an unstable seizure disorder will be excluded.
4. Females with a positive urine pregnancy test.
5. Evidence of a prior adequate trial of aripiprazole (defined as a duration of greater than or equal to 2 weeks at a dose of at least 5 mg per day). When there is not evidence of a prior adequate trial of aripiprazole, subjects must be medication-free for at least 2 weeks prior to baseline.
6. Evidence of hypersensitivity to aripiprazole (defined as an allergic response [e.g., skin rash] or potentially serious adverse effect [e.g., significant tachycardia]).
7. History of neuroleptic malignant syndrome.
8. Subjects who, in the opinion of the investigator, are unsuitable in any other way to participate in this study including being unable to comply with the requirements of the study for any reason.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2007-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Erickson, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Child and Adolescent Psychiatry Clinic - Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erickson CA, Stigler KA, Wink LK, Mullett JE, Kohn A, Posey DJ, McDougle CJ. A prospective open-label study of aripiprazole in fragile X syndrome. Psychopharmacology (Berl). 2011 Jul;216(1):85-90. doi: 10.1007/s00213-011-2194-7. Epub 2011 Feb 12. PMID 21318565

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Aripiprazole: Twelve subjects received open-label aripiprazole, mean final dose was 9.8 mg /day.
Period: Overall Study
Arm/Group | Open-label Aripiprazole
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open-label Aripiprazole: Twelve subjects received open-label aripiprazole for 12 weeks. Mean dose, 9.8 mg/day
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 14.3 [6 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 12
Aberrant Behavior Checklist [Mean (Standard Deviation); unit: units on a scale] — The Aberrant Behavior Checklist (ABC) is a 58-item measure of maladaptive behaviors and is used as a measure of drug effects. The ABC has 5 subscales: Social Withdrawal (16 items) ranging from 0 (not at all) to 48 (severe), Irritability (15 items) ranging from 0 (not at all) to 45 (severe), Inappropriate Speech (4 items) ranging from 0 (not at all) to 12 (severe), Hyperactivity (16 items) ranging from 0 (not at all) to 48 (severe), and Stereotypy (7 items) ranging from 0 (not at all) to 21 (severe). Items are rated from 0 (not at all) to 3 (severe).
  units on a scale
    ABC Irritability S | 25.3 (5.1)
    ABC Hyperactivity | 31.8 (5.8)
    ABC Social Withdrawal | 16.6 (11.8)
    ABC Stereotypy | 12.7 (5.6)
    ABC Inappropriate Speech | 6.8 (5.1)
Clinical Global Impressions - Severity [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  units on a scale | 4.5 (0.5)
Children's Yale-Brown Obsessive Compulsive Scale Modified for PDD [Mean (Standard Deviation); unit: units on a scale] — The CY-BOCS PDD has been utilized in a largescale clinical treatment study of repetitive behavior in idiopathic ASDs. CYBOCS-PDD scores range from 0 to 20 and measure repetitive/compulsive behavior and not obsessions. Higher score indicate worse outcome.
  units on a scale | 14.2 (4.6)
Social Responsiveness Scale [Mean (Standard Deviation); unit: units on a scale] — The 65-item SRS is a standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The score of each individual item is summed to create a total raw score. A total scores results are as follows: 0-62: Within normal limits 63-79: Mild range of impairment 80-108: Moderate range of impairment 109-149: Severe range of impairment
  units on a scale | 124.5 (26.7)

OUTCOME MEASURES:

1. Primary Outcome: Aberrant Behavior Checklist
Description: The Aberrant Behavior Checklist (ABC) is a 58-item measure of maladaptive behaviors and is used as a measure of drug effects. The ABC has 5 subscales: Social Withdrawal (16 items) ranging from 0 (not at all) to 48 (severe), Irritability (15 items) ranging from 0 (not at all) to 45 (severe), Inappropriate Speech (4 items) ranging from 0 (not at all) to 12 (severe), Hyperactivity (16 items) ranging from 0 (not at all) to 48 (severe), and Stereotypy (7 items) ranging from 0 (not at all) to 21 (severe). Items are rated from 0 (not at all) to 3 (severe).
Time Frame: Obtained at Baseline and Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open-label Aripiprazole: Twelve subjects received open-label aripiprazole. Mean final dose was 9.8 mg/day
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 12
units on a scale
  ABC Irritablity | 7.1 (4.4)
  ABC Hyperactivity | 15.6 (8.1)
  ABC Social Withdrawall | 9.6 (10.7)
  ABC Stereotypy | 7.6 (5.6)
  ABC Inappropriate Speech | 4.0 (3.2)

2. Primary Outcome: Clinical Global Impressions- Severity
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: Obtained at Baseline and Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 12
units on a scale | 3.5 (0.5)

3. Secondary Outcome: The Children's Yale-Brown Obsessive Compulsive Scale
Description: The CY-BOCS PDD has been utilized in a largescale clinical treatment study of repetitive behavior in idiopathic ASDs. CYBOCS-PDD scores range from 0 to 20 and measure repetitive/compulsive behavior and not obsessions. Higher score indicate worse outcome.
Time Frame: Obtained at Baseline and Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 12
units on a scale | 10.6 (5.7)

4. Secondary Outcome: Social Responsiveness Scale
Description: The 65-item SRS is a standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The score of each individual item is summed to create a total raw score. A total scores results are as follows: 0-62: Within normal limits 63-79: Mild range of impairment 80-108: Moderate range of impairment 109-149: Severe range of impairment
Time Frame: Obtained at Baseline and Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 12
units on a scale | 90.1 (31.6)

5. Secondary Outcome: The Vineland Adaptive Behavior Scales
Description: Vineland Adaptive Behavior Scales are a valid and reliable test to measure a person's adaptive level of functioning. Vineland-II forms aid in diagnosing and classifying intellectual and developmental disabilities and other disorders, such as autism spectrum disorders and developmental delays. The content and scales are organized within a 4 domain structure: Communication, Daily Living, Socialization and Motor Skills. The adaptive behavior composite standard score is computed from the sum of standard scores from the domains and converted into the adaptive behavior composite standard score. Higher scores indicate a higher adaptive level of functioning.
Time Frame: Screen Visit
Population: Data for this outcome measure are unavailable because the data file was lost during a server migration.
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 0

6. Secondary Outcome: The Vineland Maladaptive Behavior Subscales
Description: The Vineland Adaptive Behavior Scales include an optional Maladaptive Behavior Index with 27 items. The Maladaptive Behavior Index is a composite of Internalizing, Externalizing, and other types of undesirable behavior that may interfere with the individual's adaptive functioning. The Maladaptive Behavior subscale yields raw scores (0-27).
Time Frame: Week 12
Population: Data for this outcome measure are unavailable because the data file was lost during a server migration.
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Twelve Weeks
Arm/Group | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=12)
Tiredness (General disorders) | 7
Nausea/Vomiting (Gastrointestinal disorders) | 4
Drooling (General disorders) | 3
Slurred Speech (General disorders) | 2
Increased Anxiety (Psychiatric disorders) | 2
Enuresis (Renal and urinary disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Akathisia (Nervous system disorders) | 1
Increased Appetite (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No